CLINICAL TRIAL: NCT02670213
Title: A Multicentre, Non-interventional Post Marketing Study of Safety and Effectiveness of NovoThirteenR (rFXIII) During Treatment of Congenital FXIII Deficiency in Japan
Brief Title: A Study of Safety and Effectiveness of NovoThirteen® (rFXIII) During Treatment of Congenital FXIII Deficiency in Japan
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1841-4211; U1111-1162-5426 (Other: WHO)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency
MeSH Terms: interventions — recombinant factor XIII-A2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoThirteen®
  Interventions: Drug: recombinant factor XIII

INTERVENTIONS:
Drug: recombinant factor XIII — No treatment given.Patients will be treated according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
This study is conducted in Asia. Tha aim of this study is to investigate Safety and Effectiveness of NovoThirteen® (rFXIII) during treatment of congenital FXIII deficiency in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients, regardless of age, requiring treatment with NovoThirteenR for whom the treating physician has decided to use NovoThirteenR (rFXIII) treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients, regardless of age, requiring treatment with NovoThirteenR at the discretion of the treating physician
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions in patients with congenital FXIII A-subunit deficiency treated with NovoThirteen®, comprising FXIII antibodies, allergic reactions, embolic and thrombotic events and lack of therapeutic effect | Year 0-9

SECONDARY OUTCOMES:
All serious adverse events | Year 0-9
All adverse events | Year 0-9
All medical event of special interest | Year 0-9
All medication errors collected | Year 0-9
All technical complaints | Year 0-9
Use of NovoThirteen® for other uses than for the approved indication | Year 0-9
Frequency of bleeding episodes | Year 0-9

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (8):
- Japan (8):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Gamagori Hospital, Gamagori-shi, Aichi
  - Chugoku Central Hospital, Hiroshima
  - Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - Nikko Memorial Hospital, Muroran, Hokkaido,
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Takashima Municipal Hospital, Shiga
  - Ogikubo Hospital_Pediatries & Blood, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com